CLINICAL TRIAL: NCT03421691
Title: A Single-Center Open-Label Study of 1064 nm for Nonablative Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-16-EV10
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Skin Pigment; Photoaging
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Excel V laser (Other): excel V Laser Genesis procedure utilizing 1064 nm laser
  Interventions: Device: excel V Laser

INTERVENTIONS:
Device: excel V Laser — excel V Laser Genesis procedure utilizing 1064 nm laser

SUMMARY:
The purpose of this investigation is to evaluate the safety and efficacy of the Cutera excel V Laser Genesis procedure utilizing the 1064nm laser for skin rejuvenation.

DETAILED DESCRIPTION:
This is a single-center prospective, open-label uncontrolled study in 15 male or female subjects, age 35 to 55 years who desire non-ablative laser treatment for facial photo-rejuvenation, specifically improvement of rhytides, lentigines, erythema, telangiectasia and skin texture. Subjects will receive laser treatments and complete a follow up visit 12 weeks post-final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, 35 to 55 years of age (inclusive).
2. Fitzpatrick Skin Type I - IV.
3. Desires non-invasive and non-ablative treatment of skin-aging or photo-rejuvenation of the skin.
4. Have signs of moderate skin aging, including presence of mild to moderate rhytides around eyes and upper lip, multiple lentigines, diffuse erythema or telangiectasia, and a score between 4 and 7 (inclusive) on the Fitzpatrick Wrinkle Classification Scale.
5. Subject must be able to read, understand and sign the Informed Consent Form.
6. Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
7. Willing to have very limited sun exposure and use an approved sunscreen of SPF 30 or higher on the treatment area every day for the duration of the study, including the follow-up period.
8. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
9. Agree to not undergo any other procedure(s) for skin rejuvenation during the study, including but not limited to chemical peel, laser and light based device treatment, and home-use device treatment.
10. Agree to not undergo any injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler during the study.
11. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant or to father a child for the duration of the study.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser or light-based procedures or surgery.
3. Prior injection to the face of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler within 6 months of study participation, as applicable.
4. Systemic use of retinoid, such as isotretinoin, or corticosteroid, as applicable, within 6 months of study participation.
5. Use of topical medications on the face, such as antibiotics, benzoyl peroxide, retinoids (isotretinoin), corticosteroids, hydroquinone, or products containing dihydroxyacetone or alpha-hydroxy with concentration > 8%, within 1 month of participation.
6. History of malignant tumors in the target area.
7. Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
8. Pregnant and/or breastfeeding.
9. Having an infection, dermatitis or a rash in the treatment area.
10. Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
11. Suffering from coagulation disorders, or taking prescription anticoagulation medication which might make study participation unsafe according to Investigator's discretion.
12. History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
13. History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
14. History of vitiligo, eczema, or psoriasis.
15. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
16. History of seizure disorders due to light.
17. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
18. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
19. History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
20. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
21. Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
22. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
23. Current smoker or history of smoking within 6 months of study participation.
24. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

    -

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Laser and Surgery Specialists of NY and NJ, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Excel V Laser: Treatment with the excel V Laser Genesis procedure utilizing 1064 nm laser
Period: Overall Study
Arm/Group | Excel V Laser
Started | 16
Completed | 10
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Excel V Laser
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Degree of Improvement Rating at 12 Weeks Post-final Treatment
Description: The degree of improvement from Baseline observed in the post-treatment photographs at 12 weeks as assessed by independent blinded Reviewers using the Physician's Global Assessment of Improvement Scale (GAIS) Higher scores indicate better outcomes
  * 4=Very Significant Improvement
  * 3=Significant Improvement
  * 2=Moderate Improvement
  * 1=Mild Improvement 0=No Change(
Time Frame: 12 weeks post-final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Excel V Laser
Number analyzed (Participants) | 10
score on a scale | 1.4 (0.8)

ADVERSE EVENTS:
Time Frame: 12 weeks post-final treatment, up to 9 months
Arm/Group | Excel V Laser
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Excel V Laser (N=16)
Erythema (Skin and subcutaneous tissue disorders) | 16
Edema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT03421691/Prot_SAP_000.pdf